CLINICAL TRIAL: NCT06687889
Title: The Effect of Abdominal and Lumbar Muscle Stiffness Assessed by Elastography on Vertebral Fractures: A Cross-Sectional Study in Women Over 60
Brief Title: Effect of Muscle Stiffness on Vertebral Fractures in Women Over 60
Status: Completed | Type: Observational
Sponsor: Ankara City Hospital Bilkent (Other)
Collaborators: Samsun Education and Research Hospital (Other)
Responsible Party: Principal Investigator, Handan Elif Nur BAYRAKTAR, Specialist, Samsun Education and Research Hospital
Other Study IDs: Samsun-PMR-DRHENY-01
Record Dates: First submitted 2024-11-10; First posted 2024-11-14 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Osteoporosis in Post-menopausal Women; Vertebral Body Fractures; Balance, Postural
Keywords: vertebral fractures; osteoporosis; abdominal muscles
MeSH Terms: conditions — Spinal Fractures; Osteoporosis | interventions — Absorptiometry, Photon

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- vertebral fractures group: vertebral fractures group
  Interventions: Other: Elastography Measurements; Other: Bone Mineral Density Measurement (DEXA); Other: Berg balance scale; Other: Functional reach test; Other: Timed Up and Go Test
- non vertebral fractures group: non vertebral fractures group
  Interventions: Other: Elastography Measurements; Other: Bone Mineral Density Measurement (DEXA); Other: Berg balance scale; Other: Functional reach test; Other: Timed Up and Go Test

INTERVENTIONS:
Other: Elastography Measurements — Elastography Measurements
Other: Bone Mineral Density Measurement (DEXA) — Bone Mineral Density Measurement (DEXA)
Other: Berg balance scale — Berg balance scale
Other: Functional reach test — Functional reach test
Other: Timed Up and Go Test — Timed Up and Go Test

SUMMARY:
This study aims to assess the quality of lumbar and abdominal core muscles through elastography and evaluate its impact on vertebral fracture risk. This tudy's secondary objective is to investigate the relationship between muscle quality, as measured by elastography, and balance and quality of life.

The fundamental questions that this study aims to answer are as follows:

Does the quality of lumbar and abdominal core muscles, as assessed by elastography, affect the risk of vertebral fractures? Is there a relationship between muscle quality (as measured by elastography) and balance and quality of life in older adults?

DETAILED DESCRIPTION:
Osteoporosis, a systemic bone disease marked by reduced bone mass and deteriorating bone structure, increases fracture risk, especially in the spine. Vertebral fractures, most common in the lower thoracic and upper lumbar regions, can impair motor function, limit daily activities, and raise disability and mortality risks. With aging, decreasing bone mineral density (BMD) and muscle quality contribute to structural changes like kyphosis and lordosis, further reducing balance and increasing fracture risk. While DEXA remains the standard for BMD assessment, ultrasound (USG) and shear wave elastography (SWE) offer non-invasive imaging for muscle quality without radiation exposure. Despite muscle degeneration's impact on spinal stability, most osteoporosis studies focus on bones, with few examining muscles. Recognizing this gap, our study uses elastography to assess lumbar and abdominal muscle quality and its impact on vertebral fracture risk, while also exploring the relationship between muscle quality, balance, and quality of life in older adults.

ELIGIBILITY:
Inclusion Criteria:

* Female, aged ≥ 60 years

Exclusion Criteria:

* History of lumbar spine surgery
* Cancer
* Spinal infection
* Severe degenerative scoliosis
* Chronic kidney failure
* Liver cirrhosis
* Bilateral hip arthroplasty

Min Age: 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — women
Study Population: Female, aged ≥ 60 years
Sampling Method: Probability Sample
Enrollment: 81 (Actual)
Dates: Start 2024-11-24 (Actual); Primary Completion 2025-01-15 (Actual); Study Completion 2025-05-15 (Actual)

PRIMARY OUTCOMES:
Elastography Measurements | 8 weeks
  Measurements were performed using a Mindray ultrasound device (Shenzhen Mindray Biomedical Electronics Co., Ltd., Shenzhen, China) with a 15-3 MHz linear probe in Shear Wave Elastography mode. Ultrasound gel was applied between the probe and the skin to enhance contact. The probe was positioned in line with the muscle fibers and perpendicular to the skin, allowing 2D maps of each muscle's shear modulus to be obtained with a spatial resolution of 1 mm and a sampling rate of 1 sample per second. Images obtained during elastography measurements were analyzed using Q-Box to evaluate Young's modulus (kPa) and SWW (m/s). Shear modulus measurements were taken at rest and at the end of contraction. Muscle thickness measurements were recorded in mm by measuring the distance between the two fascias. All measurements were performed three times, and the average of these measurements will be used for statistical analysis

SECONDARY OUTCOMES:
Bone Mineral Density Measurement (DEXA) | 8 weeks
  All participants will undergo bone mineral density (BMD) measurements of the lumbar vertebrae (L1-L4) and left proximal femur (femur neck) at the same center using dual-energy X-ray absorptiometry (DEXA; HOLOGIC, QDR 2000, EXPLORER S1N 90910). Currently, DEXA is the standard method for diagnosing osteoporosis. Osteoporosis and osteopenia are defined according to the criteria set by the World Health Organization (WHO) for postmenopausal women: T-scores of -2.5 or lower indicate osteoporosis, while T-scores between -1.0 and -2.49 represent osteopenia. The T-score reflects bone mass by comparing it to that of a younger individual of the same sex with peak bone mass
Berg balance scale | 8 weeks
  The Berg Balance Scale is a test with proven reliability and validity in Turkish, used to assess balance in the elderly. It consists of 14 items, each scored from 0 to 4 based on observed performance. The maximum score is 56, where 0-20 points indicate balance impairment, 21-40 points suggest acceptable balance, and 41-56 points reflect good balance.
Functional Reach Test | 8 weeks
  The Functional Reach Test is a reliable and valid measure of anterior stability . The patient stands close to, but not touching, a wall with their arm extended forward at 90° flexion and fist closed. The evaluator marks the position of the third metacarpal head on the wall. The patient is then asked to reach forward as far as possible without stepping. The evaluator marks the new position of the third metacarpal head, and the difference between the initial and final marks is measured using a tape measure. Three trials are conducted, and the average is recorded. A reach of 15 cm or less indicates a significantly increased fall risk, while 15-25 cm indicates a moderate fall risk.
Timed Up and Go Test | 8 weeks
  This test, with proven reliability and validity, assesses fall risk in the elderly population. The patient is given verbal instructions to stand up from a chair, walk 3 meters following a marked line on the floor as quickly and safely as possible, turn, walk back, and sit down. Times are interpreted as follows: 10 seconds or less-patient walks independently with very low fall risk; 11-19 seconds-patient walks independently with low to moderate fall risk; 20-29 seconds-patient may occasionally need assistance, with moderate to high fall risk; over 30 seconds-patient often needs assistance and has a high fall risk.

CONTACTS AND LOCATIONS:
Locations (1):
- Samsun Education and Research Hospital, Samsun, İlkadım, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Koppenhaver SL, Scutella D, Sorrell BA, Yahalom J, Fernandez-de-Las-Penas C, Childs JD, Shaffer SW, Shinohara M. Normative parameters and anthropometric variability of lumbar muscle stiffness using ultrasound shear-wave elastography. Clin Biomech (Bristol). 2019 Feb;62:113-120. doi: 10.1016/j.clinbiomech.2019.01.010. Epub 2019 Jan 30. PMID 30721824
- [Background] MacDonald D, Wan A, McPhee M, Tucker K, Hug F. Reliability of Abdominal Muscle Stiffness Measured Using Elastography during Trunk Rehabilitation Exercises. Ultrasound Med Biol. 2016 Apr;42(4):1018-25. doi: 10.1016/j.ultrasmedbio.2015.12.002. Epub 2015 Dec 30. PMID 26746381
- [Background] Koppenhaver SL, Weaver AM, Randall TL, Hollins RJ, Young BA, Hebert JJ, Proulx L, Fernandez-de-Las-Penas C. Effect of dry needling on lumbar muscle stiffness in patients with low back pain: A double blind, randomized controlled trial using shear wave elastography. J Man Manip Ther. 2022 Jun;30(3):154-164. doi: 10.1080/10669817.2021.1977069. Epub 2021 Sep 16. PMID 34525901
- [Background] Lems WF, Paccou J, Zhang J, Fuggle NR, Chandran M, Harvey NC, Cooper C, Javaid K, Ferrari S, Akesson KE; International Osteoporosis Foundation Fracture Working Group. Vertebral fracture: epidemiology, impact and use of DXA vertebral fracture assessment in fracture liaison services. Osteoporos Int. 2021 Mar;32(3):399-411. doi: 10.1007/s00198-020-05804-3. Epub 2021 Jan 21. PMID 33475820
- [Background] Ciloglu O, Karaali E, Gorgulu FF, Ekiz T. Diaphragm thickness and stiffness in patients with hyperkyphosis due to osteoporotic vertebral fracture: an ultrasonographic and elastographic study. Pol J Radiol. 2020 Oct 5;85:e575-e580. doi: 10.5114/pjr.2020.99751. eCollection 2020. PMID 33204371
- [Background] Hug F, Tucker K, Gennisson JL, Tanter M, Nordez A. Elastography for Muscle Biomechanics: Toward the Estimation of Individual Muscle Force. Exerc Sport Sci Rev. 2015 Jul;43(3):125-33. doi: 10.1249/JES.0000000000000049. PMID 25906424
- [Background] Bedewi MA, Elsifey AA, Alfaifi T, Saleh AK, Swify SM, Sandougah KJ. Shearwave elastography of the Sartorius muscle. Medicine (Baltimore). 2021 Mar 19;100(11):e25196. doi: 10.1097/MD.0000000000025196. PMID 33726013
- [Background] Lee DG, Bae JH. Fatty infiltration of the multifidus muscle independently increases osteoporotic vertebral compression fracture risk. BMC Musculoskelet Disord. 2023 Jun 22;24(1):508. doi: 10.1186/s12891-023-06640-2. PMID 37349814
- [Background] Jeon I, Kim SW, Yu D. Paraspinal muscle fatty degeneration as a predictor of progressive vertebral collapse in osteoporotic vertebral compression fractures. Spine J. 2022 Feb;22(2):313-320. doi: 10.1016/j.spinee.2021.07.020. Epub 2021 Jul 31. PMID 34343666
- [Background] Luo Y, Yue W, Li Z, Chen L, Wang P, Sun K. An initial study of core muscles using ultrasound in postmenopausal women with osteoporosis. Ann Palliat Med. 2022 Apr;11(4):1482-1490. doi: 10.21037/apm-22-314. PMID 35523756
- [Background] Ozmen T, Gafuroglu U, Aliyeva A, Elverici E. Relationship between core stability and dynamic balance in women with postmenopausal osteoporosis. Turk J Phys Med Rehabil. 2017 Oct 6;64(3):239-245. doi: 10.5606/tftrd.2018.1674. eCollection 2018 Sep. PMID 31453517